CLINICAL TRIAL: NCT02000440
Title: Study of Losmapimod to Reduce Proteinuria in Idiopathic Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: A Phase II, Repeat Dose, Proof of Mechanism Study of Losmapimod to Reduce Proteinuria in Patients With Focal Segmental Glomerulosclerosis (FSGS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117283
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-03

CONDITIONS: Glomerulosclerosis, Focal Segmental
Keywords: GW856553; Focal segmental glomerulosclerosis (FSGS); p38 mitogen-activated protein kinase (MAPK) inhibitor; losmapimod; nephrotic syndrome
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrotic Syndrome | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Losmapimod (GW856553X) (Experimental): The subjects will be administered with 7.5 mg (1 tablet) of losmapimod following the completion of the Baseline (time zero) assessments. Subjects will continue to take one tablet in the morning and one tablet in the evening for approximately 2 weeks. After all the pre-dose assessments are completed at the Week 2 visit, subjects will be administered the first 15 mg (2 tablets) dose. Subjects will continue to take two tablets in the morning and two tablets in the evening every day for approximately 22 weeks. Doses of study treatment will be separated by at least 6 hours
  Interventions: Drug: Losmapimod

INTERVENTIONS:
Drug: Losmapimod — Losmapimod (micronized GW856553X) will be supplied as a film coated white, 7 mm round, biconvex, plain faced, tablet. Oral doses of losmapimod, 7.5 mg (1 tablet) or 15 mg (2 tablets), will be taken twice daily (BID) with food and swallowed whole (not chewed or crushed)

SUMMARY:
This is a single-arm, multicenter, open-label Phase II, proof-of-mechanism study to evaluate the efficacy, safety, tolerability and pharmacokinetics of losmapimod in approximately 21 subjects with primary (idiopathic) focal segmental glomerulosclerosis (FSGS) and substantive proteinuria as indicated by a Urinary protein/creatinine Up/c ratio >=2 gram/gram (g/g) or 24 hr urine protein >=2 g/day. Losmapimod will be orally administered twice daily over a 24-week treatment phase followed by a 12-week follow-up for safety and relapse assessments.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 70 years of age inclusive.
* Subject has a clinical diagnosis of primary (idiopathic) focal segmental glomerulosclerosis (FSGS) as verified by renal biopsy. This must be confirmed by independent review of the histopathology report and/or biopsy specimen(s) by the study central pathologist.
* Subject will have substantive proteinuria, as indicated by a spot Up/c>=2g/g or 24 hour urine total protein >=2g/day.
* A female subject is eligible to participate if she is of non-childbearing potential; criteria to be considered of 'non-childbearing potential' as described in the protocol.
* A female subject is eligible to participate if she is of child-bearing potential. Females of child-bearing potential must agree to use two of the approved contraception methods listed in the protocol from 14 days before the first dose of study drug until 30 days after the last dose of study drug. Only females of child-bearing potential with negative pregnancy test, as determined by serum human chorionic gonadotropin (hCG) test at screening and urine hCG test prior to dosing at baseline visit and during the study at the indicated times, will be administered losmapimod.
* Subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form and is willing and able to return for all study visits.

Exclusion Criteria:

* Subject has received a live attenuated vaccine within 6 weeks of first study treatment.
* Subject has collapsing FSGS lesion.
* Subject has secondary FSGS or renal impairment from a condition that is not FSGS. Causes of secondary FSGS include but are not limited to: Drugs and toxins: Analgesics, heroin, cocaine and pamidronate; Infectious or parasitic diseases: Hepatitis B, Hepatitis C, HIV (known as HIV-Associated Nephropathy), parvovirus; Adaptive structural-functional response likely mediated by glomerular hypertrophy/hyperfiltration: Hemodynamic factors - With reduced renal mass: solitary kidney, renal allograft, renal dysplasia, renal agenesis, oligomeganephronia, segmental hypoplasia, vesicoureteric reflux; Hemodynamic causes - Without reduced renal mass: sickle cell nephropathy, congenital cyanotic heart disease, hypertension; Malignancies: Lymphomas and other malignancies; for skin or cervical cancer consult medical monitor; Diabetic Nephropathy; Other forms of glomerular nephropathy: focal proliferative glomerulonephritis (IgA nephropathy, lupus, nephritis, pauci-immune focal necrotizing and crescentic glomerulonephritis), hereditary nephritis, hypertensive arterionephrosclerosis, membranous glomerulopathy, thrombotic microangiopathies; Miscellaneous: Alport syndrome, sarcoidosis, radiation nephritis; Genetic forms of FSGS (e.g. patient is known to carry FSGS causing genetic mutation).
* History of congestive heart failure.
* History of diabetes mellitus type 1 or 2.
* History of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Clinically significant systemic illness or infection within the last 28 days (e.g. chronic persistent or acute infection) that is likely to result in deterioration of the subject's condition or affect the subject's safety during the study.
* Any condition or situation, including clinically significant abnormalities in screening laboratory assessments (not related to the disease), which in the opinion of the Investigator could confound the results of the study or put the subject at undue risk.
* History of sensitivity or intolerance to the study treatment (i.e. losmapimod), or a history of drug or other allergy that in the opinion of the Investigator or GSK Medical Monitor contraindicates participation.
* Estimated GFR <45 milliliter(mL)/minutes(min)/1.73m^2 (using 4-variable Modification of Diet in Renal Disease [MDRD] formula) at screening.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >= 2xUpper Limit of Normal (ULN); alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Single QTc value obtained on the baseline ECG: QTc >=450 milliseconds (msec) (machine or manual overread); or QTc >=480 msec in subjects with Bundle Branch Block. If a single QTc is abnormal, then the averaged QTc values of triplicate electrocardiograms (ECGs) obtained (each separated by at least 5 min) will be utilized to determine eligibility.
* Hypertensive as defined as blood pressure (BP) >140/90 millimetres of mercury (mmHg) at the end of screening: If the single BP measurement is above 140 mmHg systolic or 90 mmHg diastolic, then the BP measurement can be repeated. The subject must have 2 consecutive BP readings that are less than 140 mmHg systolic and 90 mmHg diastolic, and each measurement must be separated by at least 15 minutes, to be eligible for participation in this study.
* A female subject is pregnant or nursing.
* Positive serology for chronic infection: have a historically positive Human Immunodeficiency Virus (HIV) test or test positive at screening for HIV; serologic evidence of Hepatitis B (HB) infection based on the results of testing for hepatitis B surface antigen (HBsAg), and anti- hepatitis B core antigen (HBc), positive test for Hepatitis C antibody confirmed by HCV RNA. If HCV RNA is not available, then the positive test for Hepatitis C antibody alone would be exclusionary.
* Subject having donated blood or blood products in excess of 500 mL within a 56 day period prior to the first dose of the current study.
* Participation: The subject has participated in a clinical trial where they previously received losmapimod; the subject has participated in a clinical trial and has received an investigational product 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to the first dose of the current study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07-01; Primary Completion 2016-02-29 (Actual); Study Completion 2016-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (8):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-arm, multicenter, fixed sequence open-label study consisted of 2 screening visits, run-in phase before the first dose of study treatment, followed by treatment phase in which participants received losmapimod 7.5 milligrams (mg) twice daily (BID) for 2 weeks and 15 mg BID for an additional 22 weeks, and a follow-up visit (12 weeks).
Pre-assignment Details: A total of 29 participants were screened and entered into the run-in phase, of which 17 participants received at least one dose of losmapimod.
Groups:
- Losmapimod 7.5 mg BID / 15 mg BID: Participants received losmapimod 7.5 mg BID (morning and evening), orally after 30 minutes (min.) of their starting meal for approximately 2 weeks. After all the pre-dose assessments at the Week 2 visit, participants received losmapimod 15 mg BID (2 tablets of 7.5 mg each, morning and evening), orally after 30 min. of their starting meal for approximately 22 weeks. Study treatment doses were separated by at least 6 hours.
Period: Overall Study
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Started | 17
Completed | 13
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Other-Protocol-defined Stopping Criteria | 1

BASELINE CHARACTERISTICS:
Population: Losmapimod 7.5 mg BID / 15 mg BID
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1
  Asian - Central/South Asian Heritage | 2
  Asian - East Asian Heritage | 1
  Asian - South East Asian Heritage | 2
  White - White/Caucasian/European Heritage | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting the Definition of Responder for Reduction in Proteinuria at the Indicated Time Points
Description: Proteinuria is defined as the presence of an excess of serum proteins in the urine. Participant was considered as a responder on achieving >=50 percent reduction in proteinuria from Baseline (measured as 24 hour total protein) and also having a stable renal function of >=70 percent of Baseline estimated glomerular filtration rate (eGFR) at end of treatment (>=16 Weeks). Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Week 2, Week 4, Week 8, Week 16 and Week 24
Population: Completed Treatment Population: comprised of participants who had completed >=16 weeks of losmapimod treatment or who withdrew from the treatment. Participants who withdrew prior to Week 16 were considered as non-responders.
Measure: Number; unit: Participants
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Participants
  Week 2, n= 17 | 0
  Week 4, n=15 | 1
  Week 8, n=15 | 0
  Week 16, n=13 | 0
  Week 24, n=13 | 0

2. Secondary Outcome: Number of Participants Meeting the Definition of Responder for Reduction in Proteinuria at Any Time During the Treatment Phase (Week 2 to Week 24)
Description: Proteinuria is defined as the presence of an excess of serum proteins in the urine. Participant was considered as responder on achieving >=50 percent reduction in proteinuria from Baseline (measured as 24 hour total protein) and also having a stable renal function of >=70 percent of Baseline eGFR at any time during the treatment phase of the study. Reduction in proteinuria assessment at any time during the treatment phase of the study was done by utilizing a responder analysis.
Time Frame: Any time during the treatment phase (Week 2 to Week 24)
Population: Completed Treatment Population
Measure: Number; unit: Participants
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Participants | 1

3. Secondary Outcome: Percent Change From Baseline in Urinary Protein/Creatinine (Up/c) Ratio (Spot and 24 Hours [hr])
Description: Reduction in proteinuria was measured by the Up/c ratio (spot and 24 hr) at Baseline, Week 2, 4, 8, 16, 24, end of study and at Follow-up (FU) visits Week 30 and 36. Spot urine sample was provided by the participants on site. The 24 hour urine collection started with the second morning void and ended with the first morning void on the following day; generally, 24 hour urine collection was initiated the day prior to the study visit. Baseline was defined as the value obtained at Week 0. Percent change from Baseline was calculated as change from Baseline value divided by Baseline value multiplied by 100. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 8, Week 16, Week 24, End of study, Week 30 and Week 36
Population: All Subject Population: all eligible participants who received at least one dose of investigational drug.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Percent change
  Up/c ratio 24 hr, Week 2, n= 17 | -0.45807 (25.696890)
  Up/c ratio 24 hr, Week 4, n= 15 | -0.07037 (28.954312)
  Up/c ratio 24 hr, Week 8, n= 15 | 24.32547 (39.925052)
  Up/c ratio 24 hr, Week 16, n= 13 | -10.57111 (37.211084)
  Up/c ratio 24 hr, Week 24, n= 13 | -0.59030 (29.616932)
  Up/c ratio 24 hr, End of study, n= 4 | 10.79660 (54.170928)
  Up/c ratio 24 hr, Follow-up Week 36, n= 16 | -6.56589 (43.863442)
  Up/c ratio spot, Week 2, n= 17 | 8.45052 (27.531444)
  Up/c ratio spot, Week 4, n= 16 | 11.44257 (24.783744)
  Up/c ratio spot, Week 8, n= 15 | 41.43955 (50.144228)
  Up/c ratio spot, Week 16, n= 13 | -0.99691 (34.890578)
  Up/c ratio spot, Week 24, n= 12 | 4.05899 (40.301958)
  Up/c ratio spot, End of study, n= 4 | 13.88998 (57.089949)
  Up/c ratio spot, Follow-up Week 30, n= 15 | 3.66036 (35.011255)
  Up/c ratio spot, Follow-up Week 36, n= 17 | -2.91757 (44.251282)

4. Secondary Outcome: Number of Participants With Complete Proteinuria Remissions at the Indicated Time Points
Description: Incidence of complete remissions at any time point was defined as 24 hour total protein <0.3 gram (g) per Day and maintenance of >=70 percent of Baseline eGFR throughout the treatment period. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Week 2, Week 4, Week 8, Week 16 and Week 24
Population: Completed Treatment Population
Measure: Number; unit: Participants
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Participants
  Week 2, n= 17 | 0
  Week 4, n= 15 | 0
  Week 8, n= 15 | 0
  Week 16, n= 13 | 0
  Week 24, n= 13 | 0

5. Secondary Outcome: Number of Participants Having Any Adverse Events (AEs), Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinaemia were categorized as SAE. Participants having any AE or SAE were included in the analysis.
Time Frame: From start of the study treatment (Week 0) until the Follow-up phase (Week 36)
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Participants
  Non-serious AEs | 16
  SAEs | 0

6. Secondary Outcome: Number of Participants Withdrawn Due to Toxicities
Description: Participants were monitored from start of the study treatment (Week 0) up to Week 36 for development of toxicity. Participants who developed toxicity during the period were to be withdrawn from the study.
Time Frame: From start of the study treatment (Week 0) until the Follow-up phase (Week 36)
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Participants | 0

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured in a sitting position after 5 minutes rest with comfortably seated, legs uncrossed and the back and arm supported, such that the middle of the cuff on the upper arm is at the level of the right atrium and asked to remove all clothing that covered the location of cuff placement. It was recorded at Screening, Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, End of study, and until the follow-up visit (Week 30 and Week 36). Vital sign measurements were repeated if the values were < 80 mmHg or > 140 mmHg SBP and <40 mmHg or >90 mmHg for DBP. Baseline was defined as the value obtained on Week 0. Change from Baseline was calculated as visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 8, Week 16, Week 24, End of study, and until the follow-up visit (Week 30 and Week 36)
Population: All Subject Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Millimeter of mercury (mmHg)
  SBP, Week 2, n= 17 | 3.5 (9.87)
  SBP, Week 4, n= 16 | 0.9 (12.15)
  SBP, Week 8, n= 15 | 2.0 (13.50)
  SBP, Week 16, n= 13 | -1.8 (13.16)
  SBP, Week 24, n= 13 | -1.4 (16.44)
  SBP, End of study, n=4 | 11.3 (9.00)
  SBP, Follow-up Week 30, n=15 | 0.5 (15.94)
  SBP, Follow-up Week 36, n=17 | 3.8 (15.64)
  DBP, Week 2, n= 17 | 1.5 (6.21)
  DBP, Week 4, n= 16 | -1.2 (7.81)
  DBP, Week 8, n= 15 | 1.7 (7.11)
  DBP, Week 16, n= 13 | -3.0 (9.87)
  DBP, Week 24, n= 13 | 0.2 (10.14)
  DBP, End of study, n=4 | 6.0 (7.16)
  DBP, Follow-up Week 30, n=15 | 1.3 (9.85)
  DBP, Follow-up Week 36, n=17 | 3.8 (11.84)

8. Secondary Outcome: Change From Baseline in Heart Rate at Indicated Time Points
Description: Heart rate was measured at screening, Baseline and throughout the treatment phase (Week 24) and Follow-up phase (Week 36). Heart rate measurement was repeated if the values are calculated <50 beats per minute. (bpm) or >110 bpm after the start of dosing. Baseline was defined as the value obtained at Week 0. Change from Baseline was calculated as visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 7
Population: All Subject Population
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
bpm
  Heart rate, Week 2, n= 17 | 2.6 (7.05)
  Heart rate, Week 4, n= 16 | 4.4 (8.61)
  Heart rate, Week 8, n= 15 | 2.3 (7.45)
  Heart rate, Week 16, n= 13 | 3.8 (12.08)
  Heart rate, Week 24, n= 13 | 1.5 (8.41)
  Heart rate, End of study, n=4 | 1.3 (10.31)
  Heart rate, Follow-up Week 30, n=15 | 5.3 (10.66)
  Heart rate, Follow-up Week 36, n=17 | 3.6 (11.57)

9. Secondary Outcome: Change From Baseline in Liver Function Parameters: Alkaline Phosphatase (AP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT) at Indicated Time Points
Description: Blood samples were collected at Screening (Week -4 and -2), Baseline (Week 0) and at Weeks 2, 4, 8, 16, 24 and Follow-up (Week 30 and 36) to evaluate ALT, AST, AP and GGT. Baseline was defined as the value obtained at Week 0. Change from Baseline was calculated as visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 7
Population: All Subject Population
Measure: Mean (Standard Deviation); unit: International Units/liter (IU/L)
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
International Units/liter (IU/L)
  ALT, Week 2, n= 17 | 1.8 (4.01)
  ALT, Week 4, n= 16 | 6.7 (9.44)
  ALT, Week 8, n= 15 | 7.1 (14.54)
  ALT, Week 16, n= 13 | 2.6 (6.02)
  ALT, Week 24, n= 13 | 1.2 (5.01)
  ALT, End of study, n=4 | 1.8 (3.95)
  ALT, Follow-up Week 30, n=15 | 0.5 (5.74)
  ALT, Follow-up Week 36, n=17 | 4.3 (9.47)
  AP, Week 2, n= 17 | 0.6 (10.22)
  AP, Week 4, n= 16 | -0.8 (8.92)
  AP, Week 8, n= 15 | 3.1 (8.15)
  AP, Week 16, n= 13 | 0.2 (9.04)
  AP, Week 24, n= 13 | -0.8 (7.31)
  AP, End of study, n=4 | -8.5 (21.39)
  AP, Follow-up Week 30, n=15 | 2.5 (14.38)
  AP, Follow-up Week 36, n=17 | 2.9 (20.23)
  AST, Week 2, n= 17 | 1.2 (3.34)
  AST, Week 4, n= 16 | 6.4 (16.17)
  AST, Week 8, n= 15 | 5.8 (13.99)
  AST, Week 16, n= 13 | 2.2 (5.65)
  AST, Week 24, n= 13 | -0.3 (3.20)
  AST, End of study, n=4 | -3.8 (8.18)
  AST, Follow-up Week 30, n=15 | -0.5 (5.10)
  AST, Follow-up Week 36, n=17 | 2.0 (6.89)
  GGT, Week 2, n= 17 | -1.3 (5.87)
  GGT, Week 4, n= 16 | -2.0 (9.42)
  GGT, Week 8, n= 15 | -0.7 (13.45)
  GGT, Week 16, n= 13 | -1.6 (8.65)
  GGT, Week 24, n= 13 | -2.0 (7.68)
  GGT, End of study, n=4 | -10.0 (25.10)
  GGT, Follow-up Week 30, n=15 | -0.5 (7.75)
  GGT, Follow-up Week 36, n=17 | -0.6 (13.18)

10. Secondary Outcome: Change From Baseline in Liver Function Parameters: Direct Bilirubin and Total Bilirubin at Indicated Time Points
Description: Clinical chemistry parameters: direct bilirubin and total bilirubin were assessed at Baseline (Week 0) and at Weeks 2, 4, 8, 16 24, End of studyand Follow-up (Week 30 and 36) phase. Baseline was defined as the value obtained at Week 0. Change from Baseline was calculated as visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 7
Population: All Subject Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Micromoles per liter (umol/L)
  Direct bilirubin, Week 2, n= 17 | -0.503 (1.0053)
  Direct bilirubin, Week 4, n= 16 | -0.107 (0.9811)
  Direct bilirubin, Week 8, n= 15 | -0.684 (0.8671)
  Direct bilirubin, Week 16, n= 13 | -0.263 (0.9485)
  Direct bilirubin, Week 24, n= 13 | 0.000 (0.0000)
  Direct bilirubin, End of study, n=4 | 0.000 (1.3962)
  Direct bilirubin, Follow-up Week 30, n=15 | -0.228 (0.8830)
  Direct bilirubin, Follow-up Week 36, n=17 | 0.101 (1.2783)
  Total bilirubin, Week 2, n= 17 | 0.503 (2.4754)
  Total bilirubin, Week 4, n= 16 | 0.855 (1.5295)
  Total bilirubin, Week 8, n= 15 | 0.114 (1.5112)
  Total bilirubin, Week 16, n= 13 | 0.789 (2.2745)
  Total bilirubin, Week 24, n= 13 | 0.921 (2.9300)
  Total bilirubin, End of study, n=4 | 0.855 (2.2076)
  Total bilirubin, Follow-up Week 30, n=15 | 0.684 (2.1240)
  Total bilirubin, Follow-up Week 36, n=17 | 1.006 (2.1848)

11. Secondary Outcome: Change From Baseline in Liver Function Parameters: Albumin and Total Protein at Indicated Time Points
Description: Clinical chemistry parameters: albumin and total protein were assessed at Baseline (Week 0), at Weeks 2, 4, 8, 16, 24 and Follow up (Week 30 and 36) phase. Baseline was defined as the value obtained at Week 0. Change from Baseline was calculated as visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 7
Population: All Subject Population
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Grams per liter (g/L)
  Albumin, Week 2, n= 17 | 0.4 (2.29)
  Albumin, Week 4, n= 15 | 0.2 (3.03)
  Albumin, Week 8, n= 15 | 0.4 (4.34)
  Albumin, Week 16, n= 13 | 1.8 (3.39)
  Albumin, Week 24, n= 13 | 1.8 (3.44)
  Albumin, End of study, n=4 | -1.8 (9.64)
  Albumin, Follow-up-U Week 30, n=15 | 1.9 (4.22)
  Albumin, Follow-up Week 36, n=17 | 1.8 (4.73)
  Total protein, Week 2, n= 17 | 0.0 (2.87)
  Total protein, Week 4, n= 16 | -0.6 (3.63)
  Total protein, Week 8, n= 15 | 0.8 (6.38)
  Total protein, Week 16, n= 13 | 2.4 (5.09)
  Total protein, Week 24, n= 13 | 2.8 (4.69)
  Total protein, End of study, n=4 | -1.0 (13.14)
  Total protein, Follow-up Week 30, n=15 | 2.2 (4.04)
  Total protein, Follow-up Week 36, n=17 | 2.7 (5.58)

12. Secondary Outcome: Change From Baseline in Serum Creatinine at Indicated Time Points
Description: Serum creatinine were assessed at Baseline (Week 0), at Weeks 2, 4, 8, 16, 24 and Follow-up (Week 30 and 36) phase. Baseline was defined as the value obtained at Week 0. Change from Baseline was calculated as visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 7
Population: All Subject Population
Measure: Mean (Standard Deviation); unit: Milligram per deciliter (mg/dl)
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Milligram per deciliter (mg/dl)
  Serum creatinine, Week 2, n= 17 | 0.01294 (0.150738)
  Serum creatinine, Week 4, n= 16 | 0.04187 (0.189076)
  Serum creatinine, Week 8, n= 15 | 0.11933 (0.407387)
  Serum creatinine, Week 16, n= 13 | -0.02692 (0.167252)
  Serum creatinine, Week 24, n= 13 | -0.04538 (0.267071)
  Serum creatinine, End of study, n=4 | 0.51000 (0.703468)
  Serum creatinine, Follow-up Week 30, n=15 | -0.10000 (0.271662)
  Serum creatinine, Follow-up Week 36, n=17 | 0.00588 (0.503079)

13. Secondary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR) at Indicated Time Points
Description: eGFR was calculated by using the 4-variable Modification of Diet in Renal Disease (MDRD) at Baseline (Week 0), at Weeks 2, 4, 8, 16, 24 and Follow-up (Week 30 and 36) phase. Baseline was defined as the value obtained at Week 0. Change from Baseline was calculated as visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 7
Population: All Subject Population.
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73 square meters
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
milliliter/minute/1.73 square meters
  GFR, Week 2, n= 17 | -0.29 (8.844)
  GFR, Week 4, n= 16 | -1.87 (12.148)
  GFR, Week 8, n= 15 | -5.00 (10.522)
  GFR, Week 16, n= 13 | -3.00 (15.422)
  GFR, Week 24, n= 13 | -0.38 (17.524)
  GFR, End of study, n=4 | -7.00 (14.095)
  GFR, Follow-up Week 30, n=15 | 4.87 (19.108)
  GFR, Follow-up Week 36, n=17 | 4.24 (20.398)

14. Secondary Outcome: Percent Change From Baseline in Cystatin C at Indicated Time Points
Description: Cystatin C was assessed at Baseline (Week 0), at Weeks 2, 4, 8, 16, 24 and Follow-up (Week 30 and 36) phase. Baseline was defined as the value obtained at Week 0. Change from Baseline was calculated as visit value minus value at Baseline.
Time Frame: as for outcome 7
Population: All Subject Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 17
Percent change
  Cystatin C, Week 2, n= 17 | -6.15 (13.548)
  Cystatin C, Week 4, N= 16 | -4.44 (18.610)
  Cystatin C, Week 8, n= 15 | 2.93 (17.083)
  Cystatin C, Week 16, n= 13 | -1.10 (17.267)
  Cystatin C, Week 24, n= 13 | -3.42 (19.061)
  Cystatin C, End of study, n=4 | 24.70 (47.357)
  Cystatin C, Follow-up Week 36, n=17 | 0.03 (28.071)

15. Secondary Outcome: Area Under Concentration-time Curve (AUC) From Time Zero to Time t (AUC[0-t]) and AUC From Time Zero to the End of Dosing Period (AUC[0-tau]) of Losmapimod 7.5 mg in Plasma
Description: Pharmacokinetics (PK) of losmapimod 7.5 mg was evaluated in participants with focal segmental glomerulosclerosis (FSGS) using AUC over the dosing interval of losmapimod 7.5 mg. PK samples were collected at Week 0 (pre-dose and 1, 2, 4, 6 hrs post-dose). Plasma concentration-time data were collected only up to 6 hours post the first 7.5 mg dose and only up to 2 hours post the first 15 mg dose and were not adequate to conduct a noncompartmental analysis to compare with historical data.
Time Frame: Week 0 (Pre-dose and 1, 2, 4, 6 hrs post-dose)
Population: PK Population: All participants from whom a PK sample obtained and analyzed, included in the PK population.
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 0

16. Secondary Outcome: (AUC[0-tau]) of Losmapimod 15 mg in Plasma
Description: PK of losmapimod 15 mg was evaluated in participants with FSGS using AUC over the dosing interval of losmapimod 15 mg. PK samples were collected at Week 2 (Pre-dose, 2 hrs post-dose) and Week 4, 8, 16, 24 (one of the following post-dose times: 0-2 hrs, 2-4 hrs, 4-6 hrs, and 6-8 hrs post-dose). Plasma concentration-time data were collected only up to 6 hours post the first 7.5 mg dose and only up to 2 hours post the first 15 mg dose and were not adequate to conduct a noncompartmental analysis to compare with historical data.
Time Frame: Week 2 (Pre-dose, 2 hrs post-dose) and Week 4, 8, 16, 24 (at one of the following post-dose times: 0-2 hrs, 2-4 hrs, 4-6 hrs, and 6-8 hrs post-dose)
Population: PK Population.
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 0

17. Secondary Outcome: Plasma Losmapimod 7.5 mg Maximum Observed Concentration (Cmax)
Description: PK of losmapimod 7.5 mg was evaluated in participants with FSGS using Cmax PK samples were collected at Week 0 (pre-dose and 1, 2, 4, 6 hrs post-dose). Plasma concentration-time data were collected only up to 6 hours post the first 7.5 mg dose and only up to 2 hours post the first 15 mg dose and were not adequate to conduct a noncompartmental analysis to compare with historical data.
Time Frame: Week 0 (Pre-dose and 1, 2, 4, 6 hrs post-dose)
Population: PK Population.
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of the study treatment (Week 0) until the Follow-up phase (Week 36).
Description: All Subject Population
Arm/Group | Losmapimod 7.5 mg BID / 15 mg BID
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 16/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 7.5 mg BID / 15 mg BID (N=17)
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Dizziness postural (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Fatigue (General disorders) | 4
Oedema peripheral (General disorders) | 2
Chest discomfort (General disorders) | 1
Localised oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Swelling (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Blood creatinine increased (Investigations) | 3
Blood pressure increased (Investigations) | 2
Blood albumin increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Cystatin C increased (Investigations) | 1
Eosinophils urine (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Multiple allergies (Immune system disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast pain (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.